CLINICAL TRIAL: NCT05933434
Title: Allogenic Mesenchymal Stem Cell Intraarticular Injection for Knee Osteoarthritis Therapy, an RCT Explorative Mode-of-action Study
Brief Title: Allogenic Mesenchymal Stem Cell Intraarticular Injection for Knee Osteoarthritis Therapy
Acronym: STEMJOINT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Roost Aabling, MD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STEMJOINT01
Record Dates: First submitted 2023-06-05; First posted 2023-07-06 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
Keywords: allogenic adipose derived mesenchymal stem cells; adipose derived mesenchymal stem cells; mesenchymal stem cells; stem cells
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Interventional group
  * Single intraarticular knee injection with allogenic adipose derived mesenchymal stem cells Placebo group
  * Single intraarticular knee injection with saline
Who Masked: Participant, Investigator
Masking Description: Double-blinded (participant and investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Single intraarticular knee injection with allogenic adipose derived mesenchymal stem cells (AD-MSC)
  20 million AD-MSC in 10 mL saline
  Interventions: Biological: Allogenic adipose derived mesenchymal stem cells (AD-MSC)
- Control (Placebo Comparator): Single intraarticular knee injection with saline alone
  10 mL saline
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Allogenic adipose derived mesenchymal stem cells (AD-MSC) — Laboratory isolated, cultivated and cryopreserved allogenic adipose derived mesenchymal stem cells (AD-MSC) from health donors undergoing cometic plastic surgery will be thawed on the injection day and formulated in 10 mL saline. The AD-MSCs will then be intraarticular injected using ultrasonic guidance.
  Arms: Intervention
Other: Saline — 10 mL saline will be intraarticular injected using ultrasonic guidance.
  Arms: Control

SUMMARY:
This phase I and II double blinded randomized clinical controlled trial investigates the safety and efficacy of intraarticular knee injection with allogenic adipose derived mesenchymal stem cells (AD-MSC), in patients suffering from mild-moderate knee osteoarthritis compared to placebo injection with saline.

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain (defined for at least 6 months with NRS 4 or above when pain worst)
* Patients with Grade II-III osteoarthritis according to the Kellgren Lawrence Classification and a joint width space of 1-3 mm.
* Axial hip, knee, ankle x-ray with no more than 5 degrees valgus/varus deformity
* Medial, lateral or dual compartment OA as determined above
* BMI <35
* Danish speaker
* Patients must be legally competent and must be able to sign the written consent

Exclusion Criteria:

* Severe Osteoarthritis (Grade IV according to Kellgren Lavrence Classification)
* Intraarticular tumor, infection or fracture
* Pregnancy and breast feeding
* Cognitive impairment
* Treatment with cytostatic drugs
* Previous intraarticular knee injection in the past 3 mo.
* Unable to perform MRI scan (non-compatible implants, claustrophobia and severe obesity(>BMI 35)
* Previous ligament reconstruction
* Meniscal operation with resection with more than 50% or multiple meniscal operations (more than one resection)
* Diabetes mellitus type 1 and 2
* Knee instability on physical examination
* History of allergy to antibiotics
* Concomitant severe infection, malignant tumor, coagulation diseases or uncontrolled or unmanaged systemic disease
* Presence of other types of inflammatory arthritis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Observation (change) of adverse events | Baseline, 3 months, 12 months, 24 months, 3 years, 4 years, 5 years
  Pain Diary first 30 days after treatment, any reported adverse events after treatment
Change in Knee symptoms (questionnaire Knee injury and Osteoarthritis Outcome Score (KOOS) (symptoms)) from baseline | Baseline, 3 months, 12 months, 24 months, 3 years, 4 years, 5 years
  (questionnaire Knee injury and Osteoarthritis Outcome Score (KOOS) (symptoms))

SECONDARY OUTCOMES:
Change in pain from baseline | Baseline, 3 months, 12 months, 24 months, 3 years, 4 years, 5 years
  Numeric Rating Scale (NRS)
Observation (change) of cartilage regeneration compared to baseline | Baseline, 3 months, 12 months, 24 months
  MRI Osteoarthritis Knee Score
Observation (change) of quantitative cartilage regeneration compared to baseline | Baseline, 3 months, 12 months, 24 months
  Quantitative MRI (unit: stress and strain and volumen cartilage)
Improvement (change) during clinical examination with range of motion compared to baseline | Baseline, 3 months, 12 months, 24 months
  Range of motion (unit: degrees)
Improvement (change) during clinical examination with Effusion tests (swelling) compared to baseline | Baseline, 3 months, 12 months, 24 months
  Effusion tests (swelling) (unit: effusion (YES/NO))
Improvement (change) during clinical examination with measurement of knee diameter (swelling) compared to baseline | Baseline, 3 months, 12 months, 24 months
  Measure knee diameter (unit: cm)
Improvement (change) during clinical examination with measurement of quadriceps muscle diameter (atrofi) compared to baseline | Baseline, 3 months, 12 months, 24 months
  Measure quadriceps muscle (unit: cm)

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Aabling, MD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No